CLINICAL TRIAL: NCT02165098
Title: A Single-Dose Study to Evaluate the Pharmacokinetic, Safety, Tolerability Profile and the Effects of Food on the Pharmacokinetics of Different Formulations of Cariprazine in Healthy Male Subjects
Brief Title: Cariprazine: Comparison of Slow- and Immediate-release Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGH-188-101; 2013-004925-99 (EudraCT Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Pharmacokinetic Profile
MeSH Terms: interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cariprazine PR tablet B (Experimental): Cariprazine prolonged release tablet B - fed
  Interventions: Drug: Cariprazine PR tablet B
- Cariprazine PR tablet A (Experimental): Cariprazine prolonged release tablet A - fed
  Interventions: Drug: Cariprazine PR tablet A
- Cariprazine capsule (Experimental): Cariprazine capsule - fasted
  Interventions: Drug: Cariprazine capsule
- Cariprazine prolonged release tablet B (Experimental): Cariprazine prolonged release tablet B - fasted
  Interventions: Drug: Cariprazine prolonged release tablet B
- Cariprazine prolonged release tablet A (Experimental): Cariprazine prolonged release tablet A - fasted
  Interventions: Drug: Cariprazine prolonged release tablet A

INTERVENTIONS:
Drug: Cariprazine prolonged release tablet A — Cariprazine prolonged release tablet A - fasted
  Arms: Cariprazine prolonged release tablet A
Drug: Cariprazine prolonged release tablet B — Cariprazine prolonged release tablet B - fasted
  Arms: Cariprazine prolonged release tablet B
Drug: Cariprazine capsule — Cariprazine capsule - fasted
  Arms: Cariprazine capsule
Drug: Cariprazine PR tablet A — Cariprazine Prolonged Release tablet A - fed
  Arms: Cariprazine PR tablet A
Drug: Cariprazine PR tablet B — Cariprazine Prolonged Release tablet B - fed
  Arms: Cariprazine PR tablet B

SUMMARY:
The investigators are doing this study to compare blood levels and side effects of cariprazine when it's taken as one of two 'slow release' tablets, or as an 'immediate release' capsule. The investigators will also find out if food affects the absorption of cariprazine into the bloodstream after a 'slow release' tablet.

DETAILED DESCRIPTION:
Comparison of blood levels and side effects of cariprazine when it's taken as one of two 'slow release' tablets, or as an 'immediate release' capsule. We'll also find out if food affects the absorption of cariprazine into the bloodstream after a 'slow release' tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males aged 18-55 years with body mass index (BMI) ≥ 18 kg/m2 and ≤ 30 kg/m2
* Have a semisupine pulse rate ≥ 40 bpm and ≤ 100 bpm during the vital sign assessment at screening and on admission (Day 1)
* Agree to use an effective method of contraception and not have their partners become pregnant throughout the study and for up to 4 months after the administration of the IMP, or have been sterilized for at least 1 year

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
C[max] | 0-672 hours
  Maximum Serum Concentration of the parent drug
AUC | 0-672 hours
  Area Under the Serum Concentration-Time Curve of the parent drug
T[max] | 0-672 hours
  Time to Reach the Maximum Serum Concentration of the parent drug

SECONDARY OUTCOMES:
Other PK parameters of the parent drug | 0-672 hours
  Elimination half-life period (t1/2), Mean Residence Time (MRT), if applicable
PK parameters of the metabolites, if applicable | 0-672 hours
  Maximum Serum Concentration (Cmax), Time to Reach the Maximum Serum Concentration (Tmax), (AUC0-t), Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC0-∞), Elimination half-life period (t1/2) and Mean Residence Time (MRT)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom